CLINICAL TRIAL: NCT02199626
Title: SECOND GENERATION COLON CAPSULE ENDOSCOPY (CCE-2) IN PEDIATRIC CROHN'S DISEASE (CD).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, SECOND GENERATION COLON CAPSULE ENDOSCOPY (CCE-2) IN PEDIATRIC CROHN'S DISEASE (CD)., Azienda Policlinico Umberto I
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCE-2 in pediatric CD
Record Dates: First submitted 2014-07-02; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Pediatric; Colon Capsule Endoscopy
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCE-2 (Experimental): Second generation of Colon capsule endoscopy in pediatric Crohn's disease
  Interventions: Device: Second generation of colon capsule endoscopy (GIVEN IMAGING)

INTERVENTIONS:
Device: Second generation of colon capsule endoscopy (GIVEN IMAGING)

SUMMARY:
This prospective pilot study of 40 pediatric patients with Crohn's Disease, that are candidates for endoscopic and imaging re-evaluation, examines the Given Diagnostic System and the second generation of colon capsule in comparison second generation of colon capsule endoscopy (CCE-2) to magnetic resonance enterography (MRE), small intestine contrast ultrasonography (SICUS) and endoscopy (upper and lower).

This study aims

1. To evaluate and compare the accuracy of CCE-2 with MRE, SICUS and endoscopy in the evaluation of pediatric Crohn's disease.
2. To evaluate the safety of CCE-2 in pediatric CD.

ELIGIBILITY:
Ages Eligible for Study: 6-18 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Inclusion criteria:

Subjects must meet one the following inclusion criteria to be eligible for enrollment into this proposed study:

* diagnosis of Crohn's Disease made at least 3 months before the enrolment;
* subject was referred for endoscopic and imaging follow-up in Crohn's Disease
* signed informed consent.

Exclusion criteria

The presence of any of the following will exclude a subject from study enrollment:

* Subject has dysphagia
* Subject has renal insufficiency
* Subject is known structuring Crohn's Disease identified by magnetic resonance enterography (MRE) or small intestine contrast ultrasonography (SICUS).
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the magnetic resonance enterography findings and clinical judgment of the investigator.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the accuracy of Second generation of Colon Capsule Endoscopy with magnetic resonance enterography, small intestine contrast ultrasonography and endoscopy in the evaluation of pediatric Crohn's disease. | 3 days
  Accuracy parameters (sensitivity, specificity, NPV, PPV) of second generation of colon capsule endoscopy compared to endoscopy, to magnetic resonance enterography and to small intestine contrast ultrasonography in evaluating disease activity in pediatric CD.
  The disease activity will be evaluated with a validated score (SES-CD) for endoscopy and imaging tool (damage-score).

SECONDARY OUTCOMES:
To evaluate the safety of second generation of colon capsule endoscopy in pediatric Crohn's disease. | two days
  Number, type and severity of adverse events with second generation of Crohn's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Gastroenterology and Liver Unit, Sapienza - University of Rome, Rome, Rome, Italy

REFERENCES:
- [Derived] Oliva S, Cucchiara S, Civitelli F, Casciani E, Di Nardo G, Hassan C, Papoff P, Cohen SA. Colon capsule endoscopy compared with other modalities in the evaluation of pediatric Crohn's disease of the small bowel and colon. Gastrointest Endosc. 2016 May;83(5):975-83. doi: 10.1016/j.gie.2015.08.070. Epub 2015 Sep 9. PMID 26363334